CLINICAL TRIAL: NCT06528327
Title: Bioactive Microstructured Anti Microbial Precoated Surface Implant Versus Non-coated Surface Implant in Type 2 Diabetic Patients in the Mandible (Controlled Clinical Trial)
Brief Title: Bioactive Microstructured Anti Microbial Precoated Surface Implant Versus Non-coated Surface Implant in Type 2 Diabetic Patients in the Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0375-01/2020
Record Dates: First submitted 2024-07-17; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Split Mouth Design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre coated surface implants (Experimental)
  Interventions: Other: Pre coated impants
- Non coated surface implants (Active Comparator)
  Interventions: Other: Non coated implant surface

INTERVENTIONS:
Other: Pre coated impants — Pre coated impants with microstructured bioactive antimicrobial coating with double threading for higher bone-to-implant contact and faster bone gathering on the surface.
  Arms: Pre coated surface implants
Other: Non coated implant surface — Non-coated implant with double threading for higher bone-to-implant contact and faster bone gathering on the surface.
  Arms: Non coated surface implants

SUMMARY:
Dental implant's surface properties significantly influence both biological and mechanical integration. Surface bio-treatment could accelerate and enhance bone regeneration, ensuring successful implantation. therefore, this study compares bone densification, primary and secondary stability, wound healing, and pain intensity between pre-coated antimicrobial surfaces of dental implants versus non-coated surfaces in controlled type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adequate interproximal space.
* Adequate interocclusal space.
* Adequate anatomical location, accessibility, and visualization for easy surgical implant placement.
* Both genders.
* Controlled medical condition

Exclusion Criteria:

* Presence of parafunctional dependency as bruxism.
* Adjacent pathosis near the implant site.
* Patient under radiotherapy targeting the head and neck.
* Heavy smokers.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
change in implant stability | up to 4 months
  implant stability will be assessed using Osstell device
change in pain intensity | 1st,3rd, and 7th days
  pain was assessed using visual analogue scale that ranges from 0 (No pain) to 10 (untolerated pain)
Wound Healing score | 1st,3rd, and 7th days,14th day
  Landry healing index was used;
  1. Very poor Tissue color: ≥50% of gingiva red, Response to palpation: Bleeding, Granulation tissue:Present, Incision margin: Not epithelialized, with loss ofepithelium beyond incision margin, Suppuration: Present
  2. Poor Tissue color: ≥50% of gingiva red, Response to palpation: Bleeding, Granulation tissue: Present, Incision margin: Not epithelialized, with connective tissue exposed
  3. Good Tissue colour: ≥25% and<50% of gingiva red, Response to palpation: No bleeding, Granulation tissue: None, Incision margin: No connective tissue exposed
  4. Very good Tissue colour: <25% of gingiva red, Response to palpation: No bleeding, Granulation tissue: None, Incision margin: No connective tissue exposed
  5. Excellent Tissue color: All tissues pink, Response to palpation: No bleeding, Granulation tissue: None, Incision margin: No connective tissue expose

SECONDARY OUTCOMES:
Post operative complications | 6 months
  Occurence of infection was assessed
Change in bone density | up to 4 months
  CBCT was used to measure bone density

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt